CLINICAL TRIAL: NCT04435496
Title: Study to Evaluate the Learning Curve to Anchor a Frameless Copper-releasing Device (GYN-CS®) During Caesarean Section With a Follow-up of 3 Years Study
Brief Title: Study to Evaluate the Learning Curve to Anchor GYN-CS® Device
Acronym: GYN-CS-106
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-07362
Record Dates: First submitted 2020-05-11; First posted 2020-06-17 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Learning Curve; Caesarean Section; Intra-uterine Device

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 20 healthy women between 18 and 48 years scheduled for elective Caesarean section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GYN-CS insertion (Other): GYN-CS device will be inserted in women during their c-section. The study patient can chose between a lifespan of 3 years (GYN-CS 3) and a lifespan of 10 years (GYN-CS 10) of the device.
  Interventions: Device: GYN-CS

INTERVENTIONS:
Device: GYN-CS — placement of the GYN-CS device

SUMMARY:
GYN-CS® is a new concept in intrauterine device technology. It is fixed to the uterine fundus, is frameless and entirely flexible. The GYN-CS® 3 has a lifespan of 3 years and GYN-CS® 10 has lifespan of 10 years, both used in this study. The primary objectives are: Analyse the learning curve of the surgeon and the ease of insertion of the device.

DETAILED DESCRIPTION:
This study is a mono-center, open-label, single-arm (non-randomized trial, in which each participant receives GYN-CS® 3 or GYN-CS® 10) prospective study for the insertion evaluation of GYN-CS®. Providing no complications occur, the women will remain in the study for 3 years.

The study will be conducted in 20 healthy women between 18 and 48 years scheduled for elective Caesarean section.

The learning curve parameters are the time of the procedure (starts after removal of the placenta when the uterus is completely empty and ends when the device is correctly inserted) and a scale for the ease of insertion of the device.

Following insertion of GYN-CS® 3 and 10, women will be reexamined at discharge, at 6-8 weeks, at 1, 2 and 3 years after insertion. At 3 years after insertion of the GYN-CS® 3, it will be removed during the follow-up visit. At 3 years after insertion of the GYN-CS® 10, the device doesn't need to be removed at the follow-up visit. During every visit a vaginal ultrasound and gynecological examination are performed as well as a satisfactory scale of the IUD is questioned at the patient.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, women,
* Pregnant women in the second trimester
* 18-48 years of age
* Birth by Caesarean section planned
* Be willing to stay in the study for 3 years
* Return for follow-up at the designated times
* Signed informed consent

Exclusion Criteria:

* The presence of infection of the uterus, clinical cervicitis or vaginitis (infection should be ruled out)
* Suspicion of endometrial or uterine pathology such as congenital malformation of the uterus
* Large uterine fibromata (> 3 cm in diameter)
* Acute leukemia
* Severe blood clotting disorders and undiagnosed genital tract bleeding
* Significant medical disease that in the medical opinion of the investigator is likely to interfere with patient ability to complete the entire trial
* Participants receiving corticosteroid therapy (hydrocortisone>40mg/d or an equivalent) or immunosuppressive drugs
* Caesarean section < 36 weeks

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Analyse the learning curve of the placement of the IUD by the surgeon | During the placement of the IUD
  procedure time: the time of the device placement starts after removal of the placenta when the uterus is completely empty and ends when the device is correctly inserted
Analyse the learning curve of the placement of the IUD by the surgeon | During the placement of the IUD
  successful insertion with adequate position during follow-up evaluations. The adequate position of the IUD will be checked by visualisation of the IUD by performing a vaginal ultrasound.
Ease of insertion of the IUD | During the placement of the IUD
  The ease of insertion of the IUD will be measured, using the following scale:
  * 1. The insertion of the device went smoothly
  * 2. I had little trouble inserting the device, but experienced this as a not important delay in my surgical act
  * 3. The insertion of the device was rather difficult
  * 4. The insertion of the device was time consuming, difficult and dangerous
  * 5. The insertion of the device wasn't possible due to technical issues or medical reasons

SECONDARY OUTCOMES:
Safety of insertion | During the insertion of the device until the end of the procedure of IUD placement
  All complications during the insertion of the IUD will be saved in a log
Expulsion rate and causes | During the whole duration of the trial (from the insertion of the IUD until 3 years of follow-up)
  At every follow-up visit, expulsion of the IUD will be asked and the reason will be described in a log.
Continuation rate | during the whole duration of the trial (from the insertion of the IUD until 3 years of follow-up)
  What is the reason for drop-out of the study?
Patient satisfaction: Likert scale | at every follow-up visit during the trial (4 days after the insertion of the IUD, 6-8 weeks after placement, 1 year after placement, 2 years after placement, 3 years after placement of the IUD)
  Patient satisfaction by Likert scale at every follow up: very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied or very dissatisfied. At removal, the ease of this action by the following scale for the physicians:
  * 1. I had little trouble with removing the device, but experienced this as a not important delay in my surgical act
  * 2. The removal of the device went smoothly
  * 3. The removal of the device was rather difficult
  * 4. The removal of the device was time consuming, difficult and dangerous
  * 5. The removal of the device wasn't possible due to technical issues or medical reasons
Ease if removal of the IUD | at every follow-up visite (4 days after the insertion of the IUD, 6-8 weeks after placement, 1 year after placement, 2 years after placement, 3 years after placement of the IUD)
  At removal, the ease of this action by the following scale for the physicians:
  * 1. I had little trouble with removing the device, but experienced this as a not important delay in my surgical act
  * 2. The removal of the device went smoothly
  * 3. The removal of the device was rather difficult
  * 4. The removal of the device was time consuming, difficult and dangerous
  * 5. The removal of the device wasn't possible due to technical issues or medical reasons
The pain of the patient during removal of the IUD: VAS scale | 3 years after insertion of the IUD
  The pain will be measured using a VAS scale (1. no pain, 2. mild pain, 3. nasty pain, 4. severe pain, 5. unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Kristien Roelens, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No